CLINICAL TRIAL: NCT01324115
Title: A Phase I Trial of NG-Nitro-L-Arginine (L-NNA), a Nitric Oxide Synthase Inhibitor, Given as a Single Intravenous Infusion Over 10 Minutes in Patients With Advanced Solid Tumors
Brief Title: NG-Nitro-L-Arginine in Treating Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000697500; CRUK-CR0709-11; EUDRACT-2009-013621-42
Record Dates: First submitted 2011-03-25; First posted 2011-03-28 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Nitroarginine

INTERVENTIONS:
Drug: NG-nitro-L-arginine
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: computed tomography
Procedure: dynamic contrast-enhanced magnetic resonance imaging

SUMMARY:
RATIONALE: NG-nitro-L-arginine may stop the growth of tumor cells by disrupting blood flow to the tumor.

PURPOSE: This phase I trial is studying the side effects and best dose of NG-nitro-L-arginine in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if there is a differential effect of NG-nitro-L-arginine (L-NNA) on tumor and normal tissue vasculature (blood flow/volume) in patients with advanced solid tumors in order to propose a safe recommended dose range for further evaluation.

Secondary

* To determine the correlation between plasma concentration of L-NNA and toxicity and vascular effects.
* To further determine the effects of nitric oxide synthase (NOS) inhibition on tumor tissue vasculature.
* To determine the pharmacokinetics of L-NNA.
* To determine the safety profile of L-NNA.

Tertiary

* To evaluate the potential pharmacodynamic effect of NOS inhibition on angiogenesis.
* To evaluate the effect of L-NNA on circulating NOS levels.
* To evaluate the correlation between expression levels of iNOS and eNOS and vasoconstrictive effects of L-NNA in tumor tissue (where available).

OUTLINE: This is a dose-escalation study.

Patients receive a single dose of NG-nitro-L-arginine (L-NNA) IV over 10 minutes on day 1. All patients undergo up to 6 dynamic contrast-enhanced computed tomography (DCE-CT).

Patients enrolled in the expanded cohort study undergo 4 additional scans of dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) as well as DCE-CT scans.

Blood samples are collected periodically for pharmacokinetic and biomarker studies. Samples are analyzed for L-NNA levels via a reverse-phase high performance liquid chromatography, NOS inhibition via cGMP analysis, and VEGF-A and osteopontin levels. Previously collected biopsy samples are analyzed for iNOS and eNOS expression.

After completion of study treatment and one week assessments, patients are followed up once a week for 28 days and then monthly thereafter (if required).

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced solid tumor

  * Refractory to conventional treatment or for which no conventional therapy exists or therapy is declined by the patient
* Disease assessable by DCE-CT

  * Must be a minimum size of 2 cm measured on the longest axis
* Disease assessable by DCE-MRI (patients enrolled in the expanded cohort study only)

  * Must be in sites that do not move with respiration or vascular pulsation unless this can be compensated for
* No squamous cell carcinomas

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy ≥ 12 weeks
* Hemoglobin ≥ 10.0 g/dL
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT/AST ≤ 2.5 times ULN (≤ 5 times ULN if due to tumor)
* Glomerular filtration rate ≥ 50 mL/min (uncorrected) assessed by ^51Cr-EDTA
* INR ≤ 1.4 sec
* Serum potassium normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of highly effective contraception (1 for men) 4 weeks prior to, during, and for 6 months after completion of study therapy
* No post-radiation bowel symptoms of any grade following radiotherapy within the abdomen or pelvis
* No high medical risk due to non-malignant systemic disease, including active uncontrolled infection
* No known serologically positive hepatitis B or C or HIV
* No previous or suspected allergy to imaging contrast medium
* No heart disease, including any of the following:

  * History of angina (including Prinzmetal angina) or myocardial infarction (including pathological Q waves on 12-lead ECG )
  * History of heart failure
  * History of hemodynamically significant arrhythmia (not including atrial fibrillation with well-controlled ventricular rate)
  * Cardiomyopathy (including hypertrophic cardiomyopathy, dilated cardiomyopathy, or arrhythmogenic right ventricular cardiomyopathy)
  * Hemodynamically significant valvular abnormalities (including aortic valve stenosis)
  * Congenital heart disease
* LVEF ≥ 50% by ECHO or MUGA scan
* No QT prolongation (QTc ≥ 470 msec for women and ≥ 450 for men) or any other clinically significant ECG abnormality
* No peripheral arterial disease (including all diseases caused by obstruction of large arteries in arms and legs, abdominal aortic aneurism, previous aortic dissection, or connective tissue disease resulting in thoracic aortic dilation, such as Marfan syndrome)
* No current hypertension, defined as BP consistently greater than 140/90 mm Hg or the requirement for anti-hypertensive drug treatment
* No history of thromboembolic disease or platelet/clotting disorders
* No history of cerebrovascular disease (e.g., transient ischemic attack or stroke)
* No clinically significant history of renal or hepatic impairment
* No diabetes mellitus
* Able to tolerate and comply with imaging protocol (patients with high levels of pain, urinary incontinence, or claustrophobia should be excluded)
* No other condition which, in the investigator's opinion, would not make the patient a good candidate for the clinical trial
* No pacemakers or implantable cardioverter defibrillators (for patients enrolled in the expanded cohort study only)
* No metal fragments in the eyes, shrapnel, or bullet injuries (for patients enrolled in the expanded cohort study only)

PRIOR CONCURRENT THERAPY:

* Recovered from all previous toxicities (except for alopecia or certain Grade 1 toxicities that, in the opinion of the investigator and the Drug Development Office, should not exclude the patient)
* At least 6 weeks since prior endocrine therapy

  * Stable therapy allowed if there has been no changes to the therapy within six weeks prior to treatment with L-NNA
* At least 6 weeks since prior major surgery (for patients enrolled in the expanded cohort study only)
* At least 4 weeks since prior radiotherapy (except for control of bone pain outside of the investigation site for CT evaluation), immunotherapy, or chemotherapy (6 weeks for nitrosoureas and mitomycin C)
* No prior heart or brain surgery (for patients enrolled in the expanded cohort study only)
* No major thoracic or abdominal surgery from which the patient has not yet recovered
* No concurrent drugs known to affect vascular tone (e.g., angiotensin-converting enzyme inhibitors or nitrates)
* No concurrent anticoagulants (1 mg warfarin for central line maintenance is acceptable during the trial) or anti-hypertensives
* At least 72 hours since prior non-steroidal anti-inflammatory drugs (NSAIDs), including cyclooxygenase 2 (COX2) inhibitors
* No concurrent participation or plan to participate in another interventional clinical trial

  * Participation in an observational trial is acceptable
* At least 14 days since prior and no concurrent medicines known to prolong QTc, including domperidone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) and/or subsequent maximum dose
Dose at which there is no additional differential effect of L-NNA on the tumor vasculature as measured by dynamic contrast-enhanced computed tomography (DCE-CT)
Pharmacokinetic (predominantly AUC-dependent specific vascular effects) dependent effects (duration and magnitude of effect on blood flow/volume) in the tumor tissue compared to renal tissue using data from volumetric assessments via DCE-CT

SECONDARY OUTCOMES:
Effect on tumor blood perfusion using dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) with additional blood oxygen level-dependent (BOLD) imaging and diffusion-weighted imaging (DWI) sequences
Causality of each adverse event to L-NNA and severity grade according to NCI CTCAE Version 4.02
Tertiary Outcome(s) - Measurement of L-NNA concentrations in plasma samples
Measurement of serum biomarker concentrations, osteopontin, and vascular endothelial growth factor (VEGF-A)
Measurement of NOS concentrations in circulating blood (cyclic guanine monophosphate analysis)
Measurement of iNOS and eNOS expression levels in pre-treatment tumor biopsy samples (where available)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Hoskin, MD, Principal Investigator — Mount Vernon Cancer Centre at Mount Vernon Hospital
Locations (1):
- Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England, United Kingdom